CLINICAL TRIAL: NCT07228299
Title: Supporting Families in the ICU: The Chaplain Family Project Multicenter RCT
Brief Title: Supporting Families in the ICU
Acronym: SF-ICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); Regenstrief Institute, Inc. (Other); University of California, San Francisco (Other); Wake Forest University (Other); Rush University (Other)
Responsible Party: Principal Investigator, Alexia M. Torke, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 27922; R56AG086388 (NIH)
Record Dates: First submitted 2025-10-08; First posted 2025-11-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Well-Being; Satisfaction
Keywords: spirituality; religion; surrogate decision making; proxy decision making; chaplain
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (SCAI Framework) (Experimental): Participants in this arm will receive the chaplain led intervention of the Spiritual Care Assessment and Intervention (SCAI) framework.
  Interventions: Behavioral: Spiritual Care Assessment and Intervention (SCAI) Framework
- Control (ICU Guide) (Active Comparator): Participants in this arm will participate in meetings with a member of the research team to review an ICU guide.
  Interventions: Behavioral: ICU Guide

INTERVENTIONS:
Behavioral: Spiritual Care Assessment and Intervention (SCAI) Framework — The SCAI intervention includes three visits generally scheduled 48-72 hours apart. After three visits, the chaplain will contact the surrogate at least weekly for the remainder of the hospitalization. If the patient dies, the chaplain will conduct a bereavement visit.
  The SCAI framework addresses four dimensions of spirituality. If all four dimensions are not addressed, they may be assessed during follow-up visits. If all four dimensions are addressed during the initial visit, other visits include at least one question from any dimension.
  The SCAI framework includes a list of common spiritual care interventions developed based on clinical experience and literature review.. Based on our conceptual framework, interventions are either are emotionally supportive, address spiritual or religious dimensions of care, or address information support such as exploring the meaning of medical events. Consistent with chaplain standards, the chaplain selects and tailors these interventions.
  Arms: Intervention (SCAI Framework)
Behavioral: ICU Guide — The ICU Guide intervention will include three visits with the site RA that are similar in duration to the chaplain visits (based on the single center study, first visit median of 23 minutes, follow-up visit median 12 minutes), with review of a brochure introducing the family member to the ICU including staff, policies and procedures that will be helpful to the family member.
  Arms: Control (ICU Guide)

SUMMARY:
The overarching goal of our work is to test the effect of high-quality spiritual care for ICU family surrogates on outcomes of psychological and spiritual well-being and medical decision making. Our team has developed an approach to high quality spiritual care intervention for ICU surrogates, called the Spiritual Care Assessment and Intervention (SCAI) framework, which is delivered by a chaplain interventionist to ICU surrogates.

DETAILED DESCRIPTION:
To prepare for a fully powered, multi-center study, we propose a 2-arm, attention controlled, randomized pilot trial of high-quality spiritual care for 64 surrogates at 2 additional US medical centers.

Specific Aims are:

1. To determine the feasibility and acceptability of all aspects of the study, including enrollment, randomization, delivery of the SCAI framework (e.g., chaplain intervention) and attention control conditions, acceptability, and outcome assessments, in preparation for a larger, Stage III effectiveness trial.
2. To test the effects of spiritual care on the primary outcome of anxiety (GAD-7) and the secondary outcomes of surrogate spiritual well-being and satisfaction with spiritual care (FACIT-Sp-non-illness version, Satisfaction with Care-Chaplain), and decision making for the patient, including the process of decision making and the medical care received by the patient.
3. To study the experience of spiritual care from the perspective of surrogates who are religious and those who are not, those of different faiths, and those who describe themselves as spiritual but not religious.

Because chaplains are common in the ICU this intervention is highly scalable. Results will guide hospital leaders, policy makers and the healthcare team regarding how to deploy chaplains to improve surrogates' psychological and spiritual health and the quality of decisions for critically ill patients.

ELIGIBILITY:
We will enroll patient/surrogate dyads.

Patients will be eligible if:

* They are age 18 or older at the time of screening.
* They are judged to lack decisional capacity based on either:

a Glasgow Coma Scale (GCS) score of 8 or less; or a GCS of 9-13 with at least one secondary criterion (intubation, sedation, delirium, or noted by clinicians to be unresponsive, comatose or unable to follow commands).

* They have an eligible surrogate willing to participate.

Surrogates will be eligible if:

* They are age 18 or older,
* They are considered the legally authorized representative (LAR) based on prior appointment by the patient or each state's medical consent law.

Patient/surrogate dyads will be ineligible if:

* They are unable to complete enrollment activities within 96 hours of admission to the ICU.

Patients will be ineligible if:

* They are being discharged from the ICU within 24 hours.
* They are intubated for surgery but expected to be extubated soon (typically within 24 hours).
* They are imminently dying or have a planned terminal wean.

Surrogates will be ineligible if:

*They are unable to complete study procedures in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Effect of the intervention on surrogate anxiety (GAD-7) | Assessed at baseline and 6-8 weeks after the patient has discharged from the hospital
  Generalized Anxiety Disorder- 7 (GAD-7) (7 item inventory of anxiety)- assesses subject's self-reported anxiety for the last two weeks. Scores range from 0-21 0= 'Not at all'; 1= 'Several Days'; 2= 'More than half the days'; 3= 'Nearly every day' Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for GAD.

SECONDARY OUTCOMES:
Effect of the intervention on surrogate spiritual well-being (FACIT-Sp) | Assessed at baseline and 6-8 weeks after the patient has discharged from the hospital
  Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT- Sp) Scale, a 12-item questionnaire used to measure spiritual well-being in people with chronic illnesses. It assesses aspects like meaning, peace, and faith, and is widely used in research and clinical settings, particularly for patients with cancer and other serious health conditions.
Decision making quality (FS-ICU) | Assessed 6-8 weeks after the patient has discharged from the hospital
  Family Satisfaction with the ICU Process of Decision Making Subscale, a 4 item inventory of decision making quality
Satisfaction with Spiritual Care (PSI-C) | Assessed 6-8 weeks after the patient has discharged from the hospital
  Patient Satisfaction Instrument- Chaplaincy includes 23 clinical statements which are rated on a 4 (strongly agree) to 1 (strongly disagree) scale.

OTHER OUTCOMES:
Hospice enrollment | Assessed 3 months after the patient has discharged from the hospital
  Total count of patients in both groups who enroll in hospice during the hospitalization
ICU length of stay | Assessed 3 months after the patient has discharged from the hospital
  Total length of stay for patients in both groups
DNR declaration | Assessed 3 months after the patient has discharged from the hospital
  Total count of patients in both groups who changed their code status to DNR during the hospitalization
Comfort plan initiation | Assessed 3 months after the patient has discharged from the hospital
  Total count of patients in both groups who initiated a comfort plan during the hospitalization
Receipt of life sustaining interventions | Assessed 3 months after the patient has discharged from the hospital
  Total count of patients in both groups who received life sustaining interventions during the hospitalization.
Overall distress (Distress thermometer) during the ICU stay | Days 2, 4, and 6 after enrollment and two days weekly thereafter until discharge from the ICU, up to 10 weeks.
  Total scores on distress thermometer (single item survey) will be tracked throughout the ICU stay.
Spiritual well being during the ICU stay | Days 2, 4, and 6 after enrollment and two days weekly thereafter until discharge from the ICU, up to 10 weeks.
  Spiritual well being will be assessed using the at peace single item question of spiritual distress
Decision making quality during the ICU stay for participants who make a medical decision | Days 2, 4, and 6 after enrollment and weekly thereafter until discharge from the ICU, up to 10 weeks, for those who endorse making a medical decision.
  Decision making quality scores will be based on responses to the Decisional Conflict Scale (DCS) Effective Decisions Subscale, a validated four item survey of medical decision making quality in the hospital. Scores range from 0 to 4 on each item. Scores range from 0 to 16. Higher scores indicate better decision quality. The DCS Text prompts using HIPAA compliant Twilio software will be sent.
Depression (PHQ-2) during the ICU stay | Days 1, 3, 5, and 7 after enrollment and weekly thereafter until discharge from the ICU, up to 10 weeks.
  Depression scores will be assessed using the validated 2-item version of the Patient Health Questionnaire-2. Scores range from 0 to 3 for each item. Total scores range from 0 to 6. Higher scores indicate higher likelihood of depression. Text prompts using HIPAA compliant Twilio software will be sent.
Anxiety (GAD-2) during the ICU stay | Days 1, 3, 5, and 7 after enrollment and weekly thereafter until discharge from the ICU, up to 10 weeks.
  Anxiety scores will be assessed using the validated 2-item version of the Generalized Anxiety Disorder-2. Scores range from 0 to 3 for each item. Total scores range from 0 to 6. Higher scores indicate higher likelihood of anxiety. Text prompts using HIPAA compliant Twilio software will be sent.
Communication quality (FICS-5) during the ICU stay | Days 1, 3, 5, and 7 after enrollment and weekly thereafter until discharge from the ICU, up to 10 weeks.
  Communication quality scores will be based on responses to the Family Inpatient Communication Survey-5, a validated five item survey of communication quality in the hospital. Scores range from 1 to 5 for each item. Total scores range from 5 to 25. Higher scores indicate better communication quality in the hospital. Text prompts using HIPAA compliant Twilio software will be sent.
Acceptability of the Intervention (AIM) | Assessed 6-8 weeks after the patient has discharged from the hospital
  The acceptability of the intervention measure (AIM) is a 4 item scale. Scores range from 1 to 5 for each item. Total scores range from 4 to 20. Higher scores indicate greater acceptability of the intervention.
Acceptability of psychological interventions (TAAS) | Assessed 6-8 weeks after the patient has discharged from the hospital
  The Treatment Acceptability and Adherence Scale (TAAS) is a 10 item scale developed to measure the acceptability of psychological interventions. Scores range from 1 to 7 for each item. Total scores range from 10 to 70. Higher scores indicate greater treatment acceptability and adherence.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California- San Francisco, San Francisco, California
  - Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No